CLINICAL TRIAL: NCT06273644
Title: Clinical Research on Acute Intermittent Porphyria and the Use of Carbohydrate-Rich Diet as a Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: University of Oslo (Other); Nord University (Other); UiT The Arctic University of Norway (Other); Norwegian University of Science and Technology (Other); The University of Texas Medical Branch, Galveston (Other); Karolinska University Hospital (Other); Norrlands Universitetssjukhus, Umea, Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HNF1719-24
Record Dates: First submitted 2024-02-08; First posted 2024-02-22 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Porphyria, Acute Intermittent
MeSH Terms: conditions — Porphyria, Acute Intermittent | interventions — Carbohydrates

STUDY DESIGN:
Intervention Model Description: The study is a crossover study involving 50 individuals with AIP. The study design was chosen to determine whether the treatment has an effect compared to baseline analyses and whether the sequence of treatment has an effect, as well as whether one of the interventions is more effective than the other.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding is attempted by labeling the provided diet plans as A and B. The physician recording outcome variables and the researcher performing statistical analysis are blinded to the given diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 60-65 E% Carbohydrates (Experimental): Diet plan A with 60-65 E% Carbohydrates in 4 weeks
  Interventions: Other: Carbohydrates
- 40-45% Carbohydrates (Active Comparator): Diet plan B with 40-45 E% Carbohydrates in 4 weeks
  Interventions: Other: Carbohydrates

INTERVENTIONS:
Other: Carbohydrates — Half of the patients will initially follow Diet Plan A with 60-65 E% carbohydrates for 4 weeks, followed by a 4-week washout period, and then Diet Plan B with 40-45 E% carbohydrates for 4 weeks. The other half will start with Diet Plan B for 4 weeks, followed by a 4-week washout period, and then Diet Plan A for 4 weeks . Diet Plans A and B contain recommended and adequate nutrients according to the Nordic Nutrition Recommendations 2023 (NNR2023) for maintaining a stable weight.

SUMMARY:
The main aim of this clinical trial is to learn about the effect of carbohydrate-rich diet as a treatment for AIP (acute intermittent porphyria).

Aim: Investigate the diet's impact on tissue and serum glucose, plasma insulin, cytokine levels, amino acids, and gut microbiota in AIP, and their correlation with PBG (Porphobilinogen).

Aim: Assess the diet's effect on AIP symptoms and health status in AIP. Aim: Measure the effect of a high-carbohydrate diet on mitochondrial activity in AIP Aim: Map and detect potential mutations in mitochondrial genomic DNA in AIP Aim: Discover new markers in AIP through RNA sequencing and machine learning.

Participants will follow two diet plans, a 4-week intervention with 60-65 E% carbohydrates and a 4 week intervention with 40-45 E% carbohydrates.

DETAILED DESCRIPTION:
Acute intermittent porphyria (AIP) is an inherited disease that leads to the accumulation of porphobilinogen (PBG), resulting in severe abdominal pain, paralysis, fatigue, low-grade inflammation, and an increased risk of kidney failure and liver cancer. Studies at the cellular level and in mice have shown that elevated levels of glucose and insulin can affect heme synthesis, potentially reducing PBG levels. The investigators have previously demonstrated that individuals with AIP consume less carbohydrate (E% 40) than recommended. The investigators aim to conduct a crossover study involving 50 participants with AIP, where 50% will be subjected to a 4-week intervention with 60-65 E% carbohydrates, while the other half will consume 40-45 E% carbohydrates for 4 weeks. After a 4-week intervention-free period, the two groups will switch to the respective carbohydrate percentages. Symptoms, PBG levels, continuous tissue glucose, plasma/serum insulin, glucose, cytokines, amino acid levels, microbiota in the gut, body composition, and physical activity measured using accelerometers will be assessed before and after each intervention and compared. Mitochondrial activity will be assessed at the cellular level as oxidative activity. Mutations in mitochondrial DNA and RNA will also be examined since defects in oxidative energy metabolism are known to be associated with inflammation and cancer. The work will be carried out at Nordland Hospital and at the University of Oslo. The study will be coordinated and conducted by the Postdoc and partners at Nordland Hospital, Karolinska University Hospital Stockholm and Norrland University Hospital, Umeå, the University of Oslo, the Arctic University of Tromsø, and Nord University. Clinical nutritionists will create dietary plans, and bioengineers will perform analyses. Stay abroad for postdoc, and research cooperation, with porphyria researchers at UTMB, Texas and MGH, Boston, US.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AIP

Exclusion Criteria:

* Not having diagnosis of AIP
* Undergoing treatment as part of other clinical research on AIP
* Pregnancy
* Diabetes
* Below 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-27 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Urine Porphobilinogen/creatinine | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  AIP biochemical disease activity. First morning Urine Porphobilinogen/creatinine.
  Change from baseline before diet A to immediately after diet A, and change from baseline before diet B to immediately after diet B
Urine Porphobilinogen/creatinine concentration, percentage change of repeated measurements | Day 1 ,4, 8, 11, 15, 18, 22, 25 and 29 of Diet Intervention A and of Diet Intervention B
  AIP biochemical disease activity, repeated measurements Percentage change in the median of repeated measurements of Urine Porphobilinogen/creatinine concentrations between Diet A and Diet B The repeated measurements in urine analyzed in urine samples from Day 1 ,4, 8, 11, 15, 18, 22, 25 and 29 of Diet A and of Diet B, and calculated median of Urine Porphobilinogen/creatinine concentration for diet A and median for diet B

SECONDARY OUTCOMES:
Number of Hospitalizations,sick leaves, and doctor visits due to AIP | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  Using questionnaire counting Number of hospitalizations, sick leaves, and doctor visits due to AIP
  * In the 4 weeks before Diet A, measured at baseline immediately before Diet A
  * In the 4 weeks of Diet A, measured immediately after Diet A.
  * In the 4 weeks before Diet B, measured at baseline immediately before Diet B
  * in the 4 weeks of Diet B, measured immediately after Diet B
Health status | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  A standardized questionnaire assessing health (RAND-36) with a 4-week time frame from 0 (worst functioning) to 100 (best functioning), where 2 to 5 points represent a clinically meaningful difference based on data from other chronic diseases.
Plasma Glucose level | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  Plasma glucose concentration
Interstitial fluid glucose level | Day 15 and 29 of diet A and day 15 and 29 of diet B
  Glucose measured in the interstitial fluid (ISF) Measuring is performed continuously by ISF glucose sensor FreeStyle Libre 3 in the 4 weeks of Diet A and in the 4 weeks of Diet B. Outcome is percentage change in the mean of repeated measurements between Diet A and Diet B.
  Each tissue glucose sensor lasts 14 days, and hence the outcome measure will be assessed each 14 days, and read in the LibreView program. The sensor is placed on the back of the participants upper arm
Number of hypoglycemic events | Day 15 and 29 of diet A and day 15 and 29 of diet B
  Tissue glucose measured continuously by tissue glucose sensor FreeStyle Libre 3 (Abbott) in the 4 weeks during diet A and in the 4 weeks of diet B.
  Counting number of hypoglycemic events during the 4 weeks of diet A and comparing to counted number of hypoglycemic events during the 4 weeks of diet B.
  Each tissue glucose sensor lasts 14 days, and hence the outcome measure will be assessed each 14 days, and read in the LibreView program. Assessing is performed day 15 and day 29 of diet A and day 15 and 29 of diet B.
Amino acid profile | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  Levels of amino acids measured
Plasma insulin, glucose, c-peptide | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  Concentration levels measured in plasma
HOMA score | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  HOMA score (Homeostatic Model Assessment) including estimated beta cell function, HOMA%B (%B), insulin sensitivity, HOMA%S (%S), and insulin resistance HOMA-IR (IR), calculated from insulin, glucose and C-peptide in plasma, using an Excel spreadsheet from the University of Oxford.
HbA1c | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  Concentration levels measured in blood
Cytokines in plasma | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  Cytokines, chemokines and growth factors measured using Multiplex assay from BioRad Lab, Bio-Plex 27-plex kit: Interleukin (IL)-1β, IL-1RA (IL-1 receptor antagonist), IL-2, IL-4, IL-5, IL-6, IL-7, chemokine (C-X-C) motif 8 (CXCL8), IL-9, IL-10, IL-12 (p70), IL-13, IL-15, IL-17, chemokine (C-C motif) ligand 5 (CCL5), chemokine ligand 11 (CCL11), basic fibroblast growth factor (FGF), granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), interferon (IFN)-γ, CXCL10, CCL2, CCL3, CCL4, platelet-derived growth factor-BB (PDGF-BB), tumour necrosis factor (TNF) and vascular endothelial growth factor (VEGF).
Intestinal microbiota composition | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  Sequencing of fecal samples, Gut Health Panel from Bio-Me, covering 100 different bacterias
Physical activity | Immediately after one week of Diet A, and immediately after one week of Diet B
  Accelerometer (AX3 Axivity Newcastle, UK), attached to the thigh and worn for 7 consecutive days in the first week of diet A and in the first week of diet B.
  Moderate to vigorous physical activity (MVPA) is detected in 5-second intervals. Measuring time (min/day) spent in MVPA during the first week of diet A and during the first week of diet B.
Blood pressure | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  20 min measurement
Body composition, metabolic age | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  Tanita Body Composition Analyzer
Mitochondrial oxygen consumption rate | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  SeaHorse, mononuclear cells in peripheral blood
ALAS1mRNA | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  TaqMan gene expression assay
Urine-ALA/creatinine & urine-porphyrins | Baseline before diet A and immediately after the 4 weeks of diet A, baseline before diet B and immediately after the 4 weeks of diet B
  level measurement of concentration in urine
Mitochondrial function-related genes | At baseline immediately before each participants first diet intervention
  Paxgen tubes, qPCR, Mitochondrial genome sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Elin Storjord, MD PhD, Principal Investigator — Nordlandssykehuset HF; Per Dahlqvist, MD PhD, Principal Investigator — Norrland University Hospital, Umeå; Eliane Sardh, MD PhD, Principal Investigator — Karolinska University Hospital, Stockholm
Locations (3):
- Nordland Hospital Trust, Bodø, Nordland, Norway
- Sweden (2):
  - Karolinska University Hospital, Stockholm
  - Norrland University Hospital, Umeå

IPD SHARING:
Plan to Share IPD: Yes
Selected Individual participant data that underlie the results reported in published articles, can be accessed upon reasonable request to the principal investigator, but in each case the data will be deidentified, and the data can only be shared if it is considered that it will not be possible to reidentify persons from the data, and if in each case the data protection officer has advised it and the principal investigator has granted it.
  Due to Norwegian law on sensitive data, raw data of this type cannot be submitted to public repositories, e.g DNA sequencing data.
  Study protocol and the template for informed consent form is available upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following each publication. Until 31 of December 2037
Access Criteria: Reasonable request